CLINICAL TRIAL: NCT01309438
Title: An Open-Label Study to Estimate the Effect of Multiple Doses of Erythromycin on the Pharmacokinetics, Pharmacodynamics and Safety of a Single Dose of Rivaroxaban in Subjects With Renal Impairment and Normal Renal Function
Brief Title: A Study of Erythromycin and Rivaroxaban in Study Participants With Normal and Reduced Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR017968; RIVAROXACS1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2011-02-17; First posted 2011-03-07 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Healthy; Renal Insufficiency
Keywords: Healthy; Renal Insufficiency; Rivaroxaban (BAY 59-7939, JNJ-39039039); Erythromycin; Pharmacokinetic; Pharmacodynamic
MeSH Terms: conditions — Renal Insufficiency | interventions — Rivaroxaban; Erythromycin

ARMS (3):
- Normal renal function (Experimental): Treatment Period 1 (1 dose of 10 mg rivaroxaban on Day 1) followed, up to 14 days later, by Treatment Period 2 (500 mg erythromycin three times daily on Days 1 to 6 plus 1 dose of 10 mg rivaroxaban on Day 5)
  Interventions: Drug: Rivaroxaban (normal renal function); Drug: Erythromycin (normal renal function)
- Mild renal impairment (Experimental): Treatment Period 1 (1 dose of 10 mg rivaroxaban on Day 1) followed, up to 14 days later, by Treatment Period 2 (500 mg erythromycin three times daily on Days 1 to 6 plus 1 dose of 5 mg rivaroxaban on Day 5) followed, up to 14 days later, by Treatment Period 3 (500 mg erythromycin three times daily on Days 1 to 6 plus 1 dose of 10 mg rivaroxaban on Day 5)
  Interventions: Drug: Rivaroxaban (mild and moderate renal impairment); Drug: Erythromycin (mild and moderate renal function)
- Moderate renal impairment (Experimental): Treatment Period 1 (1 dose of 10 mg rivaroxaban on Day 1) followed, up to 14 days later, by Treatment Period 2 (500 mg erythromycin three times daily on Days 1 to 6 plus 1 dose of 5 mg rivaroxaban on Day 5) followed, up to 14 days later, by Treatment Period 3 (500 mg erythromycin three times daily on Days 1 to 6 plus 1 dose of 10 mg rivaroxaban on Day 5)
  Interventions: Drug: Rivaroxaban (mild and moderate renal impairment); Drug: Erythromycin (mild and moderate renal function)

INTERVENTIONS:
Drug: Rivaroxaban (normal renal function) — One 10 mg tablet of rivaroxaban taken orally (by mouth) on Day 1 of Treatment Period 1; One 10 mg tablet of rivaroxaban taken orally on Day 5 of Treatment Period 2
  Arms: Normal renal function
Drug: Rivaroxaban (mild and moderate renal impairment) — One 10 mg tablet of rivaroxaban taken orally (by mouth) on Day 1 of Treatment Period 1; One 5 mg tablet of rivaroxaban taken orally on Day 5 of Treatment Period 2; One 10 mg tablet of rivaroxaban taken orally on Day 5 of Treatment Period 3
  Arms: Mild renal impairment; Moderate renal impairment
Drug: Erythromycin (normal renal function) — One 500 mg tablet taken orally (by mouth) three times daily on Days 1 to 6 of Treatment Period 2
  Arms: Normal renal function
Drug: Erythromycin (mild and moderate renal function) — One 500 mg tablet taken orally (by mouth) three times daily on Days 1 to 6 of Treatment Periods 2 and 3
  Arms: Mild renal impairment; Moderate renal impairment

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and pharmacodynamics of rivaroxaban when administered with erythromycin to study participants with mild or moderate renal impairment compared to the pharmacokinetics and pharmacodynamics of rivaroxaban administered to study participants with normal renal function.

DETAILED DESCRIPTION:
This is an open-label study (participants and the study physician [Investigator] will know the identity of the assigned treatments) to compare the pharmacokinetics (PK) (how the drugs are absorbed in the body) and pharmacodynamics (PD) (the actions or effects of drugs on the body) of rivaroxaban in study participants with mild or moderate renal impairment (reduced kidney function) receiving multiple doses of erythromycin, to the PK and PD of a single dose of rivaroxaban administered alone in study participants with normal renal function. The study drugs used will be rivaroxaban, a drug that acts to thin the blood to prevent the formation of blood clots, and erythromycin, an antibiotic used to treat patients with bacterial infections. Study participants with normal renal function will receive Treatment A (1 oral [by mouth] dose 10 mg rivaroxaban for 1 day) and Treatment C (500 mg oral erythromycin 3x a day (t.i.d.) on Days 1-6 + 1 oral dose of 10 mg rivaroxaban on Day 5). Study participants with mild and moderate renal impairment will receive Treatment A, Treatment B (500 mg oral erythromycin t.i.d. on Days 1-6 + 1 oral dose of 5 mg rivaroxaban Day 5), and Treatment C. Treatments A, B, and C will be separated by up to 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 38 kg/m2, inclusive
* Have a body weight of not less than 50 kg and have been characterized as having normal renal function (creatinine clearance [CLCR] > 80 mL/min), mild renal impairment (CLCR 50-79 mL/min) or moderate renal impairment (CLCR 30-49 mL/min)
* Study participants with renal impairment should have stable renal disease as determined by the Investigator

Exclusion Criteria:

* History of current clinically significant medical illness or any other illness that the Investigator considers should exclude the study participant or that could interfere with the interpretation of the study results
* Additional exclusion criteria for study participants with normal renal function include: diastolic blood pressure > 95 mm Hg and/or systolic blood pressure > 150 mm Hg)
* Additional exclusion criteria for study participants with renal impairment include: diastolic blood pressure > 100 mm Hg and/or systolic blood pressure > 170 mm Hg, other routine laboratory parameters > upper limit of normal which could not be explained by the underlying renal disease unless judged to be clinically unimportant by the investigator, have acute renal failure, or be a recipient of transplanted organs
* Have severe renal impairment (CLCR < 30 mL/min)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Rivaroxaban plasma concentrations | Up to Day 7 of Treatment Period 3
Erythromycin plasma concentrations | Up to Day 7 of Treatment Period 3
Rivaroxaban urine concentrations | Up to Day 7 of Treatment Period 3

SECONDARY OUTCOMES:
The number of patients with adverse events reported | Up to 48 hours after Day 7 of Treatment Period 3
Coagulation tests (prothrombin time [PT] and activated partial thromboplastin time [aPTT]) | Up to Day 6 of Treatment Period 3

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- United States (4):
  - Orlando, Florida
  - Minneapolis, Minnesota
  - Saint Paul, Minnesota
  - Knoxville, Tennessee

REFERENCES:
- See also: An Open-Label Study to Estimate the Effect of Multiple Doses of Erythromycin on the Pharmacokinetics, Pharmacodynamics and Safety of a Single Dose of Rivaroxaban in Subjects with Renal Impairment and Normal Renal Function — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=883&filename=CR017968_CSR.pdf